CLINICAL TRIAL: NCT01345357
Title: A Dose-Escalation Open-Label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CEP-9722 (a PARP 1 and PARP 2 Inhibitor) in Combination With Gemcitabine and Cisplatin in Patients With Advanced Solid Tumors or Mantle Cell Lymphoma
Brief Title: Study of CEP-9722 in Combination With Gemcitabine and Cisplatin in Patients With Advanced Solid Tumors or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C9722/1092; 2010-023658-36 (EudraCT Number)
Record Dates: First submitted 2011-04-19; First posted 2011-05-02 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Solid Tumors or Mantle Cell Lymphoma
Keywords: Solid tumors; mantle cell lymphoma; Gemcitabine; Cisplatin; Cancer; Neoplasms; Antineoplastic agents
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Neoplasms | interventions — CEP-9722; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEP-9722 in combination with Gemcitabine and Cisplatin (Experimental): Study drugs will be administered in cycles of 21 days for up to 6 cycles. CEP-9722 treatment will be initiated at cycle 2. After cycle 3, patients may discontinue gemcitabine and/or cisplatin for reasons of tolerability, at the discretion of the investigator.
  Interventions: Drug: CEP-9722; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: CEP-9722 — CEP-9722 will be administered orally from day 2 through day 7 of each cycle beginning with cycle 2. The starting dose will be 150 mg twice daily. Following cycle 2, the dose will either be decreased to 150 mg daily or increased to 200 mg twice daily in a cohort of 3 to 4 new patients. Subsequent cycles will increase the dose by 100 mg twice daily in cohorts of 3 to 4 patients (with criteria to expand to 6 patients) to a maximum of 400 mg twice daily. Patients must receive CEP-9722 to remain in the study. Once treatment with CEP-9722 is discontinued, patients will withdraw from the study.
Drug: Gemcitabine — Gemcitabine will be administered at 1250 mg/m^2 intravenously on day 1 and day 8 of each 21-day cycle. Dosage reduction may be applied on day 8 (within a cycle) or on day 1 of the next cycle based upon the grade of toxicity experienced by the patient.
Drug: Cisplatin — Cisplatin will be administered at 75 mg/m^2 intravenously on day 1 of each cycle, after the infusion of gemcitabine. Dosage reduction may be applied on day 1 of the next cycle based upon the grade of toxicity experienced by the patient.

SUMMARY:
The primary objective of the study is to determine the maximum tolerated dose (MTD) of CEP-9722 in combination with gemcitabine and cisplatin in patients with advanced solid tumors or mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained. The patient has a either a histologically or cytologically confirmed malignant advanced solid tumor or a mantle cell lymphoma (and has experienced failure of as least 1 previous therapy) and the patient may benefit from the combination of gemcitabine and cisplatin.
* The patient has measurable or nonmeasurable disease evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
* The patient is a man or woman at least 18 years of age.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The patient has a life expectancy of 12 weeks or more.
* The patient has adequate hematologic assessments and adequate renal and hepatic function as specified in the study protocol
* The patient has audiogram results without clinically significant abnormalities.
* The patient may have had chemotherapy provided that at least 3 weeks have elapsed and prior sequelae have resolved. If the patient has had prior radiation (curative or palliative) or prior treatment with nitrosoureas, a minimum of 4 weeks and 6 weeks, respectively, must have elapsed before treatment with CEP-9722.
* The patient has had no immunotherapy, including monoclonal antibody therapy, for at least 4 weeks and no hormonal therapy for at least 1 week, with the exception of patients with prostate cancer, who may continue hormonal therapy.
* Written informed consent is obtained.
* Agreement by women of childbearing potential (not surgically sterile or 2 years postmenopausal) to use a medically accepted method of contraception and continue the use of this method for the duration of the study and for 90 days after participation in the study. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* Agreement by men not surgically sterile or who are capable of producing offspring to practice abstinence or use a barrier method of birth control, and continue use of this method for the duration of the study and for 6 months after participation in the study.

Exclusion Criteria:

* With the exception of cancer, the patient has any serious or uncontrolled surgical, medical, or psychiatric history that could prevent compliance with study procedures, or compromise the integrity of the study.
* The patient has any of the protocol specified risk factors for Torsade de Pointes
* The patient has a brain lesion requiring systemic therapy with corticosteroids or anti-convulsive agents.
* The patient has previous hypersensitivity reactions to 1 or more of the components of the CEP-9722, gemcitabine, or cisplatin drug products.
* The patient is a pregnant or breast-feeding woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The patient is participating in another interventional clinical study at the time of enrollment or has participated in another interventional clinical study within 4 weeks prior to enrollment.
* The patient has any malabsorption syndrome and/or prior gastrectomy
* The patient has a concomitant uncontrolled and/or chronic infection or severe systemic disease.
* The patient has had previous treatment with another poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitor.
* The patient is unable to swallow tablets.
* The patient cannot interrupt continuous treatment with proton pump inhibitors and/or H2 receptor antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) of CEP-9722 in combination with gemcitabine and cisplatin in patients with advanced solid tumors or mantle cell lymphoma. | Baseline and endpoint (as soon as possible after Day 21 of the last cycle)
  To determine the maximum tolerated dose of CEP-9722, as defined by dose-limiting toxicities (DLTs) reported during the second 21-day treatment cycle (the first cycle of CEP-9722 administration).

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of CEP-9722 in combination with gemcitabine and cisplatin | During the entire study, a minimum of 6 wks (two 21-day cycles) up to a maximum of 18 wks (six 21-day cycles).
  Assessed by the occurrence of adverse events, clinical laboratory test results, vital signs measurements, electrocardiogram (ECG) findings, physical examination findings, and concomitant medication usage. Creatinine clearance will be calculated according to the Cockroft-Gault formula. An audiogram will be performed at screening and repeated during the study if clinically relevant according to the investigator. Pts who complete or withdraw from treatment will have final procedures/assessments performed as soon as possible, after day 21 of the last cycle, at the end-of-treatment visit.
Cmax pharmacokinetics parameter | Days 2 and 7 of Cycle 2 and Day 7 of Cycle 3
  To characterize the pharmacokinetics profile of CEP-8983 (the active moiety of CEP-9722) following administration of CEP-9722, through measurement of the Maximum observed drug Concentration (Cmax).
AUC pharmacokinetics parameter | Days 2 and 7 of Cycle 2 and Day 7 of Cycle 3
  To characterize the pharmacokinetics profile of CEP-8983 (the active moiety of CEP-9722) following administration of CEP-9722, through measurement of the Area Under the plasma concentration-time Curve (AUC).
Pharmacodynamics assessment | Screening and Day 2 of Cycle 2 at predose, and at 2 and 6 hours after administration of CEP-9722
  To determine the extent of poly-adenosine diphosphate ribose polymerase (PARP) inhibition in peripheral blood mononuclear cells following administration of CEP-9722
Efficacy - will be assessed by Tumor response evaluation of each patient | Screening, cycles 3 and 6, and every 2 cycles after cycle 6 until disease progression
  Tumor response will be determined using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines, when possible for patients with solid tumors. For patients with mantle tumors, tumor response may be evaluated by the International Working Group criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon, France
Locations (3):
- Teva Investigational Site 3, Brussels, Belgium
- France (2):
  - Teva Investigational Site 1, Nantes
  - Teva Investigational Site 2, Villejuif